CLINICAL TRIAL: NCT06913517
Title: Effect of Hearing Aid Versus Cochlear Implant on Hearing and Speech Recognition in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/805
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Speech Disorders
MeSH Terms: conditions — Speech Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study examines the comparative effects of hearing aids and cochlear implants on hearing and speech recognition in children with hearing loss.

This research adopts a quantitative approach to compare the outcomes of children using hearing aids versus cochlear implants. Data will be collected through audiological evaluations, including aided audiometry and speech recognition tests conducted in an audiology clinic. Descriptive and inferential statistical analyses will be used to determine differences between the groups.

DETAILED DESCRIPTION:
The study aims to provide evidence-based guidance for audiologists, educators, and caregivers regarding optimal device selection and management. By identifying the strengths and limitations of each intervention, the findings will contribute to improved rehabilitation strategies, ultimately enhancing auditory and speech outcomes in children with hearing loss. This research holds significance for advancing clinical practices in pediatric audiology.

ELIGIBILITY:
Inclusion Criteria:

* Children with 6-18 years of age
* Bilateral hearing aid users with Moderate to Severe degree Sensorineural hearing loss.
* Unilateral Cochlear Implant users with Severe to Profound degree Sensorineural hearing loss and no amplification to other ear.
* Consistent use of hearing aid or cochlear implant for more than 1 year.
* Known or presumed early onset of hearing loss before 3 years of age
* Urdu as primary language of education
* Enrolled in rehabilitation program (school or pre-school for hearing impaired children) focused on oral communication.

Exclusion Criteria:

* Children below 6 years or above 18 years
* Children with less than 1 year of consistent use of hearing aids or cochlear implant
* Children with cognitive, neurological or developmental disorders."

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study examines the comparative effects of hearing aids and cochlear implants on hearing and speech recognition in children with hearing loss.
  This research adopts a quantitative approach to compare the outcomes of children using hearing aids versus cochlear implants. Data will be collected through audiological evaluations, including aided audiometry and speech recognition tests conducted in an audiology clinic
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Aided Audiometry | 12 Months
  the hearing ability of individual using hearing aids or cochlear implant is measured in a Free Field Testing Environment using Pure Tones at frequencies 250Hz to 8000Hz.
  Interpretation: Results are plotted on Audiogram, showing the lowest level in decibel (dB HL) at which patient can detect sounds with their hearing aid or cochlear implant.
  20-30dB HL Excellent aided thresholds (satisfactory) 31-40 dBHL Mild aided thresholds (good) 41-60 dBHL Moderate aided hearing thresholds (average) More than 60dBHL Severe aided hearing thresholds (poor)
Speech Perception Test | 12 Months
  Evaluated using Phonetically Balanced Monosyllabic word list in Urdu in both quiet and noisy environment.
  Interpretation: The score is expressed as a percentage of correctly identified words under specified listening condition.
  90- 100% Normal or Slight difficulty 70-89% Mild difficulty 50-69% Moderate difficulty Below 50% Severe difficulty or poor word recognition Score

CONTACTS AND LOCATIONS:
Locations (1):
- Society for Audiological and Developmental Ailments (SADA) - Audiology Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No